CLINICAL TRIAL: NCT00857597
Title: A Randomized Controlled Trial of Transoral Incisionless Fundoplication (TIF) Versus Proton Pump Inhibitors (PPIs) for Treatment of GERD: The TIF vs. PPIs Study
Brief Title: Endoscopic Fundoplication Versus Proton Pump Inhibitors for GERD Treatment
Acronym: TvP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated after unplanned interim analysis of single centre data and results were reported
Sponsor: University of Pittsburgh (Other)
Collaborators: EndoGastric Solutions (Industry); Sandhill Scientific (Industry); Crospon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D00668-01C; PRO08110069 (Other: University of Pittsburgh)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2016-10

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; endoscopic; fundoplication; Proton Pump Inhibitors; heartburn; anti-reflux surgery
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Proton Pump Inhibitors; Esomeprazole; Omeprazole; Pantoprazole; Rabeprazole; Lansoprazole; 4-nitro-3-dimethylaminopropiophenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EsophyX (Experimental)
  Interventions: Procedure: Transoral Incisionless Fundoplication
- Proton Pump Inhibitors (Active Comparator)
  Interventions: Drug: Proton Pump Inhibitors; active control

INTERVENTIONS:
Procedure: Transoral Incisionless Fundoplication — The TIF procedure using the EsophyX system with SerosaFuse fasteners was designed to create full-thickness serosa-to-serosa plications and construct valves of 3-5 cm in length and 200-300° in circumference.
  Other Names: TIF procedure; ELF procedure; Endoluminal fundoplication; Endoscopic fundoplication
  Arms: EsophyX
Drug: Proton Pump Inhibitors; active control — Proton Pump Inhibitors; active control
  Other Names: Esomeprazole; Lansomeprazole; Omeprazole; Pantoprazole; Rabeprazole; Nexium; Prevacid; Dakar; Lanso; Lanzor; Prezal; Lanzol; Prilosec; Losec; Logastric; Protonix; Zurcal; Pantozol; Zurcale; Aciphex; Pariet
  Arms: Proton Pump Inhibitors

SUMMARY:
The study objective is to evaluate the relative merits, safety and effectiveness of Transoral Incisionless Fundoplication (TIF) in GERD patients currently treated with daily Proton Pump Inhibitors (PPIs).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Proven gastroesophageal reflux (pH < 4 for > 4.3% time while off PPIs for 7-14 days)
* On daily PPIs for > 1 year
* Recurrence of GERD symptoms (GERD-HRQL score difference of > 10 between on and off PPIs)
* Normal or hypotonic LES resting pressure (5-40 mmHg)
* Patient willingness to cooperate with random group assignment, attend 4-5 office visits and comply with all tests in this protocol
* Signed informed consent

Exclusion Criteria:

* BMI > 35
* Hiatal hernia > 2 cm
* Esophagitis grade D
* Barrett's esophagus
* Esophageal stricture
* Esophageal ulcer
* Esophageal motility disorder
* Gastric motility disorder
* Prior splenectomy
* Gastric paralysis
* Pregnancy (in females)
* Immunosuppression
* ASA > 2
* Portal hypertension
* Coagulation disorders
* Previous antireflux procedure
* Any other health condition, which the investigator believes would prevent the patient from completing the study
* Lack of fluency in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
GERD symptoms | Baseline
GERD symptoms | 6 month follow-up
GERD symptoms | 12 month follow-up

SECONDARY OUTCOMES:
PPI usage | at 0, 6 and 12 month follow- up
Lower esophageal acid exposure | at 0, 6 and 12 month follow- up
Esophagitis | at 0, 6 and 12 month follow- up
  Percentage of Participants with Esophagitis (Los Angeles classification scale)
Rate of adverse events | at 0, 6 and 12 month follow- up

CONTACTS AND LOCATIONS:
Overall Officials: Blair A Jobe, MD, Principal Investigator — University of Pittsburgh Medical Center; Nicole D Bouvy, MD, PhD, Principal Investigator — University Hospital Maastricht, The Netherlands
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- See also: Data reported in Am J Gastroenterol. 2015 Apr;110(4):531-42. doi: 10.1038/ajg.2015.28. Epub 2015 Mar 31. — https://www.ncbi.nlm.nih.gov/pubmed/25823768